CLINICAL TRIAL: NCT05939414
Title: An International, Prospective, Open-label, Multi-center, Randomized Phase III Study Comparing Lutetium (177Lu) Vipivotide Tetraxetan (AAA617) Versus Observation to Delay Castration or Disease Recurrence in Adult Male Patients With Prostate-specific Membrane Antigen (PSMA) Positive Oligometastatic Prostate Cancer (OMPC)
Brief Title: An Open-label Study Comparing Lutetium (177Lu) Vipivotide Tetraxetan Versus Observation in PSMA Positive OMPC.
Acronym: PSMA-DC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA617D12302; 2022-502956-29-00 (Other: EU CT number)
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Oligometastatic Prostate Cancer (OMPC)
Keywords: Lutetium (177Lu) vipivotide tetraxetan; Oligometastatic Prostate Cancer (OMPC); Metastasis Free Survival (MFS); gallium (68Ga) gozetotide; piflufolastat (18F); prostate-specific membrane antigen (PSMA); Delay Castration; Stereotactic Body Radiation Therapy (SBRT); metastasis-directed therapy; Androgen Deprivation Therapy (ADT)-free survival.
MeSH Terms: interventions — Lutetium-177

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational Arm: lutetium (177Lu) vipivotide tetraxetan (AAA617) (Experimental): All participants will be treated with Stereotactic Body Radiation Therapy (SBRT) to all metastatic lesions followed by a dose of 7.4 GBq (200 mCi) +/- 10% of AAA617 which will be administered once every 6 weeks (1 cycle) for a planned 4 cycles.
  Interventions: Drug: AAA617
- Control arm: observation (watchful waiting) (No Intervention): All participants will be treated with Stereotactic Body Radiation Therapy (SBRT) to all metastatic lesions followed by observation only.

INTERVENTIONS:
Drug: AAA617 — Stereotactic Body Radiation Therapy (SBRT) followed by AAA617 will be administered once every 6 weeks (1 cycle) for a planned 4 cycles to participants randomized to the Investigational arm
  Other Names: (177Lu) vipivotide tetraxetan
  Arms: Investigational Arm: lutetium (177Lu) vipivotide tetraxetan (AAA617)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of lutetium (177Lu) vipivotide tetraxetan (AAA617) in participants with oligometastatic prostate cancer (OMPC) progressing after definitive therapy to their primary tumor. The data generated from this study will provide evidence for the treatment of AAA617 in early-stage prostate cancer patients to control recurrent tumor from progressing to fatal metastatic disease while preserving quality of life by delaying treatment with androgen deprivation therapy (ADT).

DETAILED DESCRIPTION:
All participants will be assessed for eligibility and will undergo baseline disease assessments including a mandatory gallium (68Ga) gozetotide (also known as [68Ga]Ga-PSMA-11) or piflufolastat (18F) ( also known as[18F]DCFPyL) PET/CT scan and CI (i.e., CT/MRI and bone scans).

Piflufolastat (18F) PET/CT scan will be performed in countries where it is approved.

Stereotactic Body Radiation Therapy (SBRT) will be administered to all metastatic Prostate Cancer (PC) lesions after randomization and before the start of treatment with AAA617 or observation.

* The duration of SBRT procedures is approximately 3 weeks.
* For participants randomized to the investigational arm (AAA617), the treatment duration will be up to 4 cycles of AAA617. For participants randomized to the control arm (observation) the treatment duration will end at the last fraction of SBRT administration.
* The visit frequency will be every week 1 and 3 of each of the 4 cycles and every 16 weeks thereafter (for both arms) until first event of disease progression (RECIST 1.1)
* The study duration is approximately 6.5 years.

ELIGIBILITY:
Key Inclusion criteria:

1. Histologically confirmed prostate cancer prior to randomization
2. Participants must have biochemically recurrent disease after definitive treatment to prostate by Radical Prostatectomy ((RP), (alone or with post-operative radiation to prostate bed/pelvic nodes)) or External beam Radiation Therapy (EBRT), (prostate alone or prostate with seminal vesicle and/or pelvic nodes) and/or brachytherapy prior to randomization. Biochemical recurrence (BCR) is defined as: nadir PSA + 2 ng/mL post XRT (if participant received-radiation therapy to intact prostate) and PSA > 0.2 ng/mL and rising post RP (with or without post-operation Radiation Therapy (RT))
3. Participants must have OMPC with 1-5 PSMA -positive metastatic lesions on screening PSMA PET/CT scan (with either gallium (68Ga) gozetotide or piflufolastat (18F)) as visually assessed by BIRC. For definition of PSMA PET positivity, please refer to Section 8.1 and the Imaging Manual. Metastatic lesions may include regional/pelvic lymph nodes (N1), distant lymph nodes (M1a), bone (M1b), lung and others visceral (M1c) except liver and brain classified using American Joint Committee on Cancer (AJCC) 8. When counting the number of oligometastatic lesions, each lesion is counted as distinct metastasis irrespective of its anatomical location (e.g., one pelvic and one extra-pelvic lymph node will be counted as two metastatic lesions)
4. At least 1 PSMA-positive lesion must be a distant metastasis (M1) per AJCC8 classification at screening. For AJCC M staging, PSMA PET/CT information should be used
5. Participants must have a negative CI for M1 disease at screening.

   Note:
   * For a participant not to be eligible, CI positive M1 lesions should be unequivocal in CI scans, i.e., potentially not attributable to findings thought to represent something other than tumor (e.g., degenerative, or post-traumatic changes or Paget's disease in bone lesions). For CI assessments, bone lesions must be assessed by bone scan only and soft tissue lesions must be assessed by CT/MRI scans only at screening.
   * Prior knowledge of PSMA PET positivity should not influence the radiologist (reader) in determination of CI positivity. Two different readers will be involved, one reader for PSMA PET/CT scan and one reader for CI: Reader will be blinded to PSMA PET scan results while reading CI scans. Reader should not modify their assessment of CI scans (e.g. changing a lesion previously identified as equivocal in CI to unequivocal) after reading the PSMA PET scan. Similarly, biopsy positivity should not influence the reader in the assessment of CI positivity. More details on the reading paradigm will be provided in the imaging charter
   * MRI for radiation treatment planning may show M1 disease but this will not exclude the participant from the study if the lesion is deemed negative per baseline CT or bone scans
   * Participants with pelvic disease (N1) seen in CI are allowed if the local spread is below common iliac bifurcation (per AJCC 8 definition of local disease)
   * Distant lymph node disease (M1a) that is visible per CI and less than 10mm in the short axis is not exclusionary irrespective of PSMA PET positivity.
   * If a previously surgically removed lesion was unequivocal for M1 by bone scan or CT, the participant is not eligible.
6. All metastatic lesions detected at screening must be amenable to SBRT
7. Non-castration testosterone level >100 ng/dL at screening

Key Exclusion criteria:

1. Participants with de novo OMPC at screening
2. Unmanageable concurrent bladder outflow obstruction or urinary incontinence at screening. Note: participants with bladder outflow obstruction or urinary incontinence, which is manageable and controlled with best available standard of care (incl. pads, drainage) are allowed
3. Prior therapy with:

   1. ADT (including bilateral orchiectomy) and ARPIs used for metastatic prostate cancer treatment

      * Participants who received AR-directed therapy, whether ADT or an ARPI or both, as neoadjuvant or adjuvant therapy as a component of their primary therapy, are eligible provided that they discontinued therapy ≥12 months prior to randomization for ADT (i.e., 12 months after the last day of the last injection) or ≥3 months if ARPI was given as monotherapy. ARPI's as a term includes both contemporary androgen synthesis inhibitors (e.g., abiraterone, galeterone, and orteneronel), and receptor inhibitors (enzalutamide, apalutamide and darolutamide).
      * Patients who biochemically relapsed after primary therapy may also have had treatment with AR directed therapy and participants who had SBRT with ADT are also eligible provided that the ARPI +/- ADT or ADT alone was terminated

        ≥12 months prior to randomization for ADT (i.e., 12 months after the last day of the last injection) or ≥3 months if ARPI was given as monotherapy.
      * Participants who received first generation anti-androgens (bicalutamide, flutamide, nilutamide, cyproterone) for biochemical recurrence or adjuvant/neoadjuvant therapy are eligible provided that they discontinued therapy ≥3 months prior to randomization.
      * Participants who have discontinued ADT due to disease progression are not eligible (i.e., Castration-Resistant Prostate Cancer (CRPC) participants)
   2. Other hormonal therapy. e.g.,

      •Use of estrogens, 5-α reductase inhibitors (finasteride, dutasteride), other steroidogenesis inhibitors (aminoglutethimide) if used in the context of prostate cancer treatment. Same medications are allowed if used for other indications: e.g., Benign Prostatic Hyperplasia (BPH), if stopped ≥3 months before randomization.
   3. Radiopharmaceutical agents (e.g., Strontium-89, PSMA-targeted radioligand therapy)
   4. Immunotherapy (e.g., sipuleucel-T)
   5. Chemotherapy, except if administered in the adjuvant/neoadjuvant setting completed > 12 months before randomization
   6. Any other investigational or systemic agents for metastatic disease
4. Radiation therapy external beam radiation therapy (EBRT) and brachytherapy within 28 days before randomization
5. Concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, hormonal therapy (see ADT initiation guidance in Section 6.8.2), Poly Adenosine Diphosphate-Ribose Polymerase (PARP) inhibitor, biological therapy or investigational therapy
6. Diagnosed at screening with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. However, participants with a prior history of malignancy that has been adequately treated and who have been disease/treatment free for more than 3 years are eligible, as are participants with adequately treated non-melanoma skin cancer and superficial bladder cancer.
7. History or current diagnosis of ECG abnormalities indicating significant risk of safety for participants participating in the study such as:

   * Concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, and clinically significant second or third degree Atrioventricular (AV) block without a pacemaker
   * History of familial long QT syndrome or known family history of Torsades de Pointe
8. Participants in immediate need of ADT as assessed by the investigator.

Other protocol defined Inclusion/Exclusion may apply.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2028-04-25 (Estimated); Study Completion 2031-10-03 (Estimated)

PRIMARY OUTCOMES:
Blinded Independent Review Committee (BIRC) assessed Metastasis Free Survival (MFS) | From date of randomization until first evidence of radiographically detectable bone or soft tissue distant metastasis or death due to any cause, whichever occurs first, assessed up to approximately 30 months
  Blinded Independent Review Committee (BIRC) assessed Metastasis Free Survival (MFS) is defined as the time from randomization to first evidence of radiographically detectable bone or soft tissue distant metastasis by conventional imaging (i.e., Computed Tomography (CT)/Magnetic Resonance Imaging (MRI) and bone scans) as assessed by BIRC using RECIST 1.1 or death due to any cause, whichever occurs first.
  Participants who are alive without distant metastasis at the analysis data cut-off or are lost to follow-up at the time of analysis will be censored for MFS at the time of their last adequate radiographic assessment. Clinical deterioration without objective radiographic evidence will not be considered as documented distant metastasis.

SECONDARY OUTCOMES:
Key secondary endpoint: Time to Hormonal Therapy (TTHT) | From date of randomization until date of Androgen Deprivation Therapy (ADT), assessed up to approximately 74 months
  Time to Hormonal Therapy (TTHT) is defined as the time from randomization to the time to Androgen Deprivation Therapy (ADT). The type of hormonal therapy will be at the discretion of the Investigator.
Investigator assessed Metastasis Free Survival (MFS) | From date of randomization until first evidence of radiographically detectable bone or soft tissue distant metastasis or death from any cause, whichever occurs first, assessed up to approximately 74 months
  Investigator assessed Metastasis Free Survival (MFS) is defined as the time from randomization to the first evidence of radiographically detectable bone or soft tissue distant metastasis by conventional imaging (i.e., CT/MRI and bone scans) as assessed by Investigator using RECIST 1.1 or death from any cause, whichever occurs first.
Time to prostate specific antigen (PSA) progression (TTPSAP) | From date of randomization until date of first PSA progression, assessed up to approximately 74 months
  Time to prostate specific antigen (PSA) progression (TTPSAP) is defined as time from randomization to first PSA progression 1. First PSA progression 1 is defined as a rising PSA confirmed on repeated measurement at least 3 weeks later, and at least greater than 25% and >= 2 ng/mL above nadir or baseline, whichever is lower. In the absence of PSA progression, TTPSAP will be censored at the last PSA measurement.
Radiographic Progression Free Survival (rPFS) | From date of randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 74 months
  Radiographic progression free survival (rPFS) is defined as the time from randomization to first documentation of confirmed radiographic progressive disease or death due to any cause (whichever occurs first) by conventional imaging (i.e., CT/MRI and bone scans) using RECIST 1.1. The rPFS will be analyzed based on BIRC and Investigator assessments respectively.
Time to next therapy (local or systemic) | From date of randomization until initiation of the next line of therapy (local or systemic), assessed up to approximately 74 months
  Time to next therapy (local or systemic) is defined as the time from randomization to initiation of the next line of therapy (local or systemic). Next-line therapy is defined as the first new (local or systemic) anti-neoplastic therapy initiated after discontinuation of study treatment regardless of end of treatment (EOT) reason.
24-month prostate-specific antigen (PSA) progression free survival (PFS) | From date of randomization until date of first documented PSA progression 2 or death from any cause, whichever occurs first, assessed up to approximately 74 months
  24-month PSA PFS is defined as PSA PFS at 24 months. PSA PFS is defined as the time from date of randomization to the date of first documented PSA progression 2 or death from any cause, whichever occurs first. PSA progression 2 is defined as a PSA concentration above the nadir (or baseline if lower) of >= 0.5 ng/mL, confirmed by repeated measurement at least 3 weeks later. PSA PFS will be censored if no PSA PFS event is observed before the first to occur analysis cut-off date. The censoring date will be the date of the last adequate tumor assessment prior to cut-off.
Time to symptomatic progression | From date of randomization until date of first documented symptomatic progression, assessed up to approximately 74 months
  Time to symptomatic progression is defined as time from randomization to the date of first documented event for any of the following, whichever occurs first: development of symptomatic skeletal event, escalation in cancer-related pain or worsening of disease-related symptoms leading to the initiation of a new systemic anticancer therapy, development of clinically significant symptoms due to local or regional tumor progression leading to surgery or radiation therapy.
Functional Assessment of Cancer Therapy - Prostate (FACT-P) Questionnaire | From date of randomization up till 42 day safety Follow-up, assessed up to approximately 74 months
  FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS). The FACTGeneral (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
Functional Assessment of Cancer Therapy - Radionuclide Therapy (FACT-RNT) Questionnaire | From date of randomization up till 42 day safety Follow-up, assessed up to approximately 74 months
  The FACT-RNT (Functional Assessment of Cancer Therapy - Radionuclide Therapy) is a Patient Reported Outcomes (PRO) new measure developed using FACIT specific questions (items), selected from FACIT item bank, to assess treatment-related symptoms of special interest associated with radioligand therapies.
  The FACT-RNT contains items assessing dry mouth, dry eyes, vomiting, diarrhea, constipation, loss of appetite, fatigue, impact of fatigue, bone pain, and isolation due to illness or treatment. FACT-RNT score range 0 to 60, with higher score indicating better quality of life.
Brief Pain Inventory - Short Form (BPI-SF) Questionnaire | From date of randomization up till 42 day safety Follow-up, assessed up to approximately 74 months
  The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item selfreport questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression is defined as an increase in score of 30% or greater from baseline without decrease in analgesic use.
European Quality of Life (EuroQol) - 5 Domain 5 Level scale (EQ-5D- 5L) | From date of randomization up till 42 day safety Follow-up, assessed up to approximately 74 months
  EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.
Time to First Symptomatic Skeletal Event (TTSE) | From date of randomization till end of treatment (EOT) or death, whichever happens first, assessed up to approximately 74 months
  Time to first symptomatic skeletal event (TTSSE) is defined as date of randomization to the date of first new SSE or death from any cause, whichever occurs first. Symptomatic skeletal events (SSE) will be defined by the occurrence of any of the following (whichever occurs earlier): symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain.
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | From date of randomization up till 42 day safety Follow-up, assessed up to approximately 74 months
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Dose modifications and intensity for AAA617 | From date of randomization until end of treatment (EOT), assessed up to approximately 30 months
  Dose modifications (dose interruptions and reductions) and dose intensity for AAA617 will be assessed and summarized using descriptive statistics.
Overall survival (OS) | From date of randomization until date of death from any cause, assessed up to approximately 74 months
  Overall Survival (OS) is defined as the time from the date of randomization to the date of death due to any cause. OS time for participants who are alive at the end of the study or are lost to follow-up will be censored at the date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (131):
- United States (38):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - VA Greater LA Healthcare System, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University, Palo Alto, California
  - UCSF, San Francisco, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - The Cancer Institute of Alexian Brothers, Elk Grove, Illinois
  - Unity Point Clinic, Des Moines, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - East Jefferson Hospital, Metairie, Louisiana
  - University of Maryland Medical Ctr, Baltimore, Maryland
  - Johns Hopkins Kimmel Com Cancer Ctr, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - BAMF Health, Grand Rapids, Michigan
  - Profound Research LLC, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - VA St Louis Health Care System, St Louis, Missouri
  - Wash U School of Medicine, St Louis, Missouri
  - Adult and Pedi Urology and Urogyne, Omaha, Nebraska
  - Memorial Sloane Ketterin Cancer Ctr, New York, New York
  - Associated Med Professionals of NY, Syracuse, New York
  - Montefiore Hospital, The Bronx, New York
  - East Carolina University, Greenville, North Carolina
  - Dayton Physicians, Kettering, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Univ of Texas Southwest Med Center, Dallas, Texas
  - Rio Grande Urology, El Paso, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Center, Wytheville, Virginia
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Caba
- Australia (4):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Malvern, Victoria
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Wilrijk
- Novartis Investigative Site, São Paulo, São Paulo, Brazil
- Canada (7):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- China (3):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Czechia (3):
  - Novartis Investigative Site, Ostrava, Poruba
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- France (6):
  - Novartis Investigative Site, Saint-Cloud, Hauts De Seine
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Herblain
- Germany (7):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Rostock
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Hungary (2):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
- Israel (5):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Italy (8):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Negrar, VR
- Japan (9):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Fukushima
  - Novartis Investigative Site, Kyoto
- Malaysia (2):
  - Novartis Investigative Site, Petaling Jaya, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Huxquilucan
- Novartis Investigative Site, Amsterdam, Netherlands
- VA Caribbean Healthcare System, San Juan, Puerto Rico
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (4):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Trenčín
- Spain (7):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Switzerland (3):
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lucerne
  - Novartis Investigative Site, Zurich
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (5):
  - Novartis Investigative Site, Bristol, Avon
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com